CLINICAL TRIAL: NCT06007989
Title: Assessing the Relationship Between Hypoxia and the Immune Environment in Myeloma Patients (CHIME)
Acronym: CHIME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTsp212
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Myeloma
Keywords: multiplex; immunohistochemistry; hypoxia; single-cell RNA sequencing; pimonidazole; myeloma; microenvironment; metabolomics
MeSH Terms: conditions — Neoplasms, Plasma Cell; Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basic science study, no intervention.: Basic science study, no intervention.

SUMMARY:
The study is looking at how myeloma is related to low oxygen levels (hypoxia) in the bone marrow. This is to understand the disease better. It might also guide treatment in the future.

For the study, we will run tests on a portion of the samples taken during a bone marrow biopsy. A bone marrow biopsy is taken as part of the diagnosis or follow up of myeloma. The tests in our study will look closely at the make-up of immune cells in the bone marrow, highlight areas of low oxygen, and look at genetic changes in cells from low-oxygen areas. We will ask patients to take a capsule the day before their bone marrow biopsy containing pimonidazole hydrochloride, a substance which will show up areas of low oxygen on tests.

Overall we want to know:

1. If myeloma cells 'live' in areas of low oxygen in the bone marrow
2. What are the immune and bone marrow cells which are neighbours of myeloma cells?
3. Are there genetic changes in low oxygen myeloma cells

   For the pilot study, we want to know:
4. Can we use new techniques to study questions 1-3? The techniques we want to use are pimonidazole with multiplex immunohistochemistry and single cell RNA sequencing.

The information we get from the tests will help us get a better understanding of how myeloma works. Future studies may also use these results to develop new kinds of drugs for myeloma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients referred to The Christie NHS Foundation Trust from another hospital with proven multiple myeloma which may be either treatment naïve or previously treated.

  2. Aged 18 or over 3. World Health Organisation (WHO) performance status 0 to 2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks 4. Provision of written informed consent 5. Willing to undergo a bone marrow biopsy 6. Willing to take pimonidazole hydrochloride

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to staff at the study site)
2. Evidence of any significant clinical disorder or laboratory finding that made it undesirable for the patient to participate in the study
3. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with newly diagnosed or previously treated myeloma
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of the utility of a set of investigational tools for investigating the bone marrow microenvironment in myeloma patients | Assessment is at the time of diagnosis.
  Specifically we aim to determine the feasibility of using pimonidazole as a marker of hypoxia in conjunction with: A) Multiplex immunohistochemistry to characterise the spatial organization of cellular inflammatory elements and myeloma cells in the bone marrow, B)Single cell RNA sequencing to characterise the expression profile of myeloma cells in hypoxic areas of marrow

CONTACTS AND LOCATIONS:
Overall Officials: Emma Searle, MBChB, MA, MRCP, FRCPath, PhD, Principal Investigator — University of Manchester, The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient level data is unlikely to be useful to other groups in this small pilot study.